CLINICAL TRIAL: NCT02146664
Title: The Role of DLBS1033 in The Management of Acute Non-ST Elevation of Myocardial Infarction (NSTEMI) Without Early Coronary Revascularization
Brief Title: DLBS1033 for Acute NSTEMI Without Early Coronary Revascularization
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: The investigational cases were no longer relevant considering the recent implementation of our current national healthcare system.
Sponsor: Dexa Medica Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DLBS1033-0513
Record Dates: First submitted 2014-05-13; First posted 2014-05-26 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2016-04

CONDITIONS: Acute Non-ST Elevation Myocardial Infarction
Keywords: Acute NSTEMI; DLBS1033; SPECT; Infarct size; Left ventricular function
MeSH Terms: conditions — Non-ST Elevated Myocardial Infarction | interventions — DLBS 1033

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DLBS1033 (Experimental): DLBS1033 enteric-coated tablet is administered at the dose of 490 mg, one tablet three times daily, everyday for eight weeks of study period
  Interventions: Drug: DLBS1033
- Placebo (Placebo Comparator): Placebo is administered one tablet three times daily, everyday for eight weeks of study period
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DLBS1033 — Investigational drug or placebo will be given in addition to the standard therapy which consists of: aspirin enteric-coated tablet 1 x 160 mg (two tablets @ 80 mg) and clopidogrel film-coated tablet 1 x 75 mg daily for eight weeks. Standard therapy alone will still be given afterwards, for another sixteen weeks
  Other Names: Disolf
  Arms: DLBS1033
Drug: Placebo — Investigational drug or placebo will be given in addition to the standard therapy which consists of: aspirin enteric-coated tablet 1 x 160 mg (two tablets @ 80 mg) and clopidogrel film-coated tablet 1 x 75 mg daily for eight weeks. Standard therapy alone will still be given afterwards, for another sixteen weeks
  Arms: Placebo

SUMMARY:
This is a prospective, randomized, double-blind, double-dummy, and controlled study of DLBS1033 in the management of acute non-ST elevation myocardial infarction (NSTEMI) without early coronary revascularization. It is hypothesized that the combination of DLBS1033 with aspirin and clopidogrel will result in greater reduction of infarct size in comparison with that of aspirin and clopidogrel alone.

DETAILED DESCRIPTION:
After diagnosed NSTEMI, patient is hospitalized and given medications according to the standard management of acute NSTEMI, including anticoagulant low molecular weight heparin. Eligible subjects are then randomized to receive either DLBS1033 at a dose of 490 mg three times daily or its placebo in addition to clopidogrel 75 mg once daily and aspirin 160 mg once daily for an 8-week course of therapy. Afterwards, the administration of DLBS1033 and its placebo are stopped, while the dual antiplatelet therapy (aspirin and clopidogrel) remains for another 16 weeks at the same dose regimen as the previous.

Clinical and laboratory examinations to evaluate the investigational drug's efficacy and safety are performed at baseline, week 4, week 8, and week 24. To guard the safety of the study subjects, haemostasis parameters, hematology parameters, and CRUSADE bleeding score are evaluated every two-week-interval over the first eight weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Men and women of 30-75 years of age.
* Evidence of acute non-ST elevation myocardial infarction (NSTEMI) at screening, as confirmed by all of the following:

  * ECG transient ST-segment deviation/depression (≥ 1 mm) or prominent T-wave inversion, in multiple precordial leads;
  * Positive plasma biomarkers of myocardial necrosis: cardiac troponin I (cTnI);
  * Clinical symptoms of chest discomfort/pain or anginal equivalent (dyspnea, diaphoresis, excessive vomiting in diabetic patients and arm or jaw pain).
* High risk subjects, defined as having Thrombolysis in Myocardial Infarction (TIMI) score ≥ 4
* Subjects refuse to undergo reperfusion therapies, such as coronary artery-bypass surgery (CABG) or percutaneous coronary intervention (PCI) within the next six months.
* Therapy with study medication can be started within 7 days after first presentation in the hospital.
* Able to take oral medication.

Exclusion Criteria:

* For females of childbearing potential: pregnancy, breast-feeding, the intention of becoming pregnant.
* ECG presentation of STEMI.
* History of hemorrhagic stroke within the last 3 months.
* Patients with seizure at the onset of stroke or with regular medication for seizure/epilepsy.
* History of serious head injury within the last 3 months.
* History of major surgery within the last 3 months.
* Ongoing long term need for oral anticoagulants, antiplatelets, fibrinolytic, or antithrombotic agents, other than the study medication.
* Having any implanted pacemaker or cardiac resynchronization therapy (CRT) or cardiac resynchronization therapy defibrillators (CRT-D).
* Clinically significant arrhythmias or atrioventricular conduction block greater than first degree.
* Acute or chronic heart failure as defined by the New York Heart Association (NYHA) classification as functional Class IV.
* Known severe LV dysfunction (EF ≤ 40 and EDD > 55 mm).
* Inadequate liver function: ALT > 3 times upper limit of normal (ULN).
* Inadequate renal function: serum creatinine ≥ 1.5 times upper limit of normal (ULN).
* Uncontrolled hypertension (SBP > 185 mmHg or DBP > 110 mmHg).
* Random plasma glucose ≥ 180 mg/dL and HbA1c ≥ 7.0% at Screening.
* Moderate to high risk of bleeding, defined as those who have the CRUSADE bleeding score of > 30.
* Known or suspected allergy to any of study medications used in the study, including other lumbrokinase products.
* Prior experience with DLBS1033 or other oral lumbrokinase products.
* Clinical evidence of malignancies with survival period < 1 year.
* Any other disease which judged by the investigator could interfere with trial participation or trial evaluation.
* Enrolled in other interventional protocol within 30 days prior to Screening.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-11; Primary Completion 2017-11 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Infarct size | Week 0, week 8, week 24
  The quantitative change of infarct size, measured using SPECT.

SECONDARY OUTCOMES:
LV function | Week 0, week 4, week 8, and week 24
  Improvement in left ventricular (LV) function, measured by 2D echocardiography.
Composite endpoints | Week 0 - 24
  Composite endpoints (composite of major adverse cardiovascular events), comprising of all-cause of death, recurrent myocardial infarction or ischemic stroke within the study period.
Individual event of MACE and other cardiovascular events | Week 0 - 24
  Individual event of MACE and other cardiovascular events, such as: shock, pulmonary oedema, congestive heart failure, arrhythmias, hemodynamic instability/cardiogenic shock, including the presence of new infarct(s) within the study period.
Nitroglycerin amount | Week 0 - 24
  Number of nitroglycerin (rescue medicine) taken during the study period.
Plasma fibrinogen level | Week 0, 4, 8, and 24
  Change in plasma fibrinogen level.
Plasma d-dimer level | Week 0, 4, 8, and 24
  Change in plasma d-dimer level.
hs-CRP | Week 0, 4, 8, and 24
  Change in hs-CRP.
Routine hematology | Week 0, 4, 8, and 24
  Routine hematology measured includes: hemoglobin, hematocrit, RBC, WBC, differentiation of WBC, and platelet count. Particularly for hemoglobin and hematocrit level, they are measured at baseline and every interval of 2 weeks over the first 8 weeks of treatment and at the end of study (week 24).
Liver function | Week 0, 4, 8, and 24
  Liver function measured includes: serum ALT (SGPT), serum AST (SGOT), alkaline phosphatase, and total bilirubin. Particularly for serum ALT, it is measured at baseline and every interval of 2 weeks over the first 8 weeks of treatment and at the end of study (week 24).
Renal function | Week 0, 4, 8, and 24
  Renal function measured includes: serum creatinine and BUN. Particularly for serum creatinine, it is measured at baseline and every interval of 2 weeks over the first 8 weeks of treatment and at the end of study (week 24).
Haemostasis parameter | Week 0, 4, 8, and 24
  Haemostasis parameter measured includes: prothrombin time (PT), International Normalized Ratio (INR), and activated partial thromboplastin time (aPTT). Particularly for PT and INR, they are measured at baseline and every interval of 2 weeks over the first 8 weeks of treatment and at the end of study (week 24).
Adverse event | Week 0 - 24
  Adverse events (especially major and minor bleeding) are observed and carefully evaluated along the course of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Munawar, SpJP(K), MD, Principal Investigator — Binawaluya Cardiac Hospital; Ismi Purnawan, SpJP(K), MD, Principal Investigator — Central Army Hospital RSPAD Gatot Soebroto
Locations (2):
- Indonesia (2):
  - Central Army Hospital RSPAD Gatot Soebroto, Central Jakarta, Jakarta Special Capital Region
  - Binawaluya Cardiac Hospital, Jakarta, Jakarta Special Capital Region